CLINICAL TRIAL: NCT05652777
Title: Feasibility of Vital Sign Assessment by Community Health Workers During Antenatal Care Community Outreach
Brief Title: Feasibility of Using NeoSpot at Community Settings
Status: Completed | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Neopenda, PBC (Industry); Wellcome Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3109-2022
Record Dates: First submitted 2022-09-13; First posted 2022-12-15 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related
Keywords: Pregnancy; Vital signs; Wearable medical devices
MeSH Terms: interventions — Vital Signs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women attending antenatal care clinic during routine community outreach activities in Lusaka, Zambia.
  Interventions: Device: NeoSpot

INTERVENTIONS:
Device: NeoSpot — Pregnant women will undergo screening of their vital signs using the NeoSpot device.
  Other Names: Vital sign measurement

SUMMARY:
Continuous vital sign monitoring is a basic tenet of specialized care in the developed world that is vastly underutilized during hospital or clinic admissions or outpatient routine visits in most low-and-middle income countries (LMICs). Despite the positive outcomes associated with vital sign monitoring (i.e., increased survival-to-discharge rates, lower complication rates and shorter length of stay in hospital), the prohibitive costs of conventional patient monitors and the difficulty in maintaining complex medical equipment limit its practice in the developing world.

Currently, due to lack of medical supplies, most ANC clinics - within the health facilities or during outreach activities - do not monitor for vital signs and blood pressure among pregnant women. While many devices exist, their ease of use and high-cost, including maintenance costs, hinder screening and monitoring programs in low resource settings. Accurate and low-cost vital sign monitoring devices are required to improve identification and treatment of women with danger signs during their routine ANC visits. To meet the growing demand for vital sign monitors during the COVID-19 pandemic, Neopenda has adapted an affordable, wearable, wireless vital sign monitoring solution (neoSpotTM), that measures temperature, respiration rate, blood oxygen saturation, pulse rate, and blood pressure.

DETAILED DESCRIPTION:
Continuous vital sign monitoring is a basic tenet of specialized care in the developed world that is vastly underutilized during hospital or clinic admissions or outpatient routine visits in most low-and-middle income countries (LMICs). Despite the positive outcomes associated with vital sign monitoring (i.e., increased survival-to-discharge rates, lower complication rates and shorter length of stay in hospital),1 the prohibitive costs of conventional patient monitors and the difficulty in maintaining complex medical equipment limit its practice in the developing world.

Wearable health devices (WHDs) are increasingly helping people better monitor their health status both at an activity/fitness level for self-health tracking and at a medical level providing more data to healthcare providers to increase the potential for early diagnosis and guidance of treatment. Key advancements in technology are enabling the creation of smaller computers than ever before; allowing wearable technology to incorporate miniaturized systems to enhance the quality and convenience of patient care.1 Advances in materials science, chemical analysis techniques, equipment design and manufacturing methods have further laid the foundation for the continuous evolution of wearable systems over the years.2

WHDs when properly designed, implemented and adopted can provide ample benefits for healthcare providers and patients. Wearable technologies like Apple watch, Fitbit, Jawbone, ViSi Mobile and Vital Connect wireless patch have been used in tracking personal physiological and biological parameters for routine activity performance and/or clinical monitoring.3,4 These devices collect data such as heart rate, stress levels, obesity, oxygen saturation, blood pressure and calories; and serve a broad range of use cases from newborn to elderly patients in different settings such as hospitals, nursing homes and homecare settings.

Measurement of vital signs in both in- and out-patient departments and during community outreach activities is necessary to assess the clinical situation of the patient and capture early warning scores for deterioration. The currently practice in most LMICs is for a clinician to take routine vital sign measurements intermittently and manually record these on a clinical chart. However, this leaves a lot of room for missed detection of early warning scores. Delays in diagnosing clinical deterioration prevent clinicians from taking corrective actions and are associated with increased complication rates and mortality. The use of wearable devices for long term monitoring is intended to provide instant diagnosis of acute events that will in turn lead to more effective and timely treatment of patients.5 Furthermore, the situation becomes more dire during community outreach activities (i.e., child health week, community ANC outreach, etc.), which are usually conducted by limited clinicians and several community health workers (CHWs).

In contrast to the traditional monitoring devices that have been in use in clinical settings, WHDs may be more suited to the constraints of low-resources settings. Conventional medical equipment frequently fail in health facilities in LMICs due to complex design and specifications, and environmental constraints including power instability, internet access, space limitations and availability of spare parts. This calls upon the need for more feasible innovations to improve on the quality of care for people living in LMICs. WHDs offer a promising solution.

Currently, due to lack of medical supplies, most ANC clinics - within the health facilities or during outreach activities - do not monitor for vital signs and blood pressure among pregnant women. While many devices exist, their ease of use and high-cost, including maintenance costs, hinder screening and monitoring programs in low resource settings. Accurate and low-cost vital sign monitoring devices are required to improve identification and treatment of women with danger signs during their routine ANC visits. To meet the growing demand for vital sign monitors during the COVID-19 pandemic, Neopenda has adapted an affordable, wearable, wireless vital sign monitoring solution (neoSpotTM), that measures temperature, respiration rate, blood oxygen saturation, pulse rate, and blood pressure.

ELIGIBILITY:
Pregnant women:

Inclusion criteria

1. Pregnant
2. 18+ years of age
3. Willing to consent

Exclusion criteria

1. Unable to consent
2. Not pregnant
3. Age below 18 years

In-depth Interviews:

1. Community Health Workers who have used the NeoSpot device
2. Pregnant women who have experienced the device and enrolled in the study

2. 18+ years of age 3. Willing to consent

Exclusion criteria

1. Pregnant women not enrolled in the study
2. Unable to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women residing at Kanyama compound and attending ANC care during routine community outreach activities will be approached, screened, and consented for study participation.
  Community Health Workers who have used the device on enrolled study participants (pregnant women) will under-go in-depth interviews.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a wearable, wireless vital sign monitoring solution NeoSpot device by Community Health Workers (CHWs) | Baseline to day 1
  To describe the feasibility of CHWs to use the NeoSpot device during community ANC outreach through in-depth interviews
Acceptability of using a wearable, wireless vital sign monitoring solution NeoSpot device by Community Health Workers (CHWs) | Baseline to day 1
  To describe the acceptability of CHWs to use the NeoSpot device during community ANC outreach through in-depth interviews

SECONDARY OUTCOMES:
Acceptability of using a wearable, wireless vital sign monitoring solution NeoSpot device by pregnant women | Baseline to day 1
  To describe the acceptability of pregnant women to be screened using the NeoSpot device during community ANC outreach through in-depth interviews
Collect photoplethysmograph (PPG) data using a wearable, wireless vital sign monitoring solution NeoSpot device | Baseline to day 1
  To obtain raw PPG data from the prototype NeoSpot device which will be used in the development of an accurate and reliable blood pressure algorithm.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Manasyan, MD, Principal Investigator — Center for Infectious Disease Research in Zambia (CIDRZ)
Locations (1):
- Kanyama First Level Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be available to other researchers upon reasonable request to the study PI.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: Following study closure and publication of the main study findings.
Access Criteria: De-identified study data will be available to other researchers upon reasonable request to the study PI.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT05652777/Prot_SAP_000.pdf